CLINICAL TRIAL: NCT02974322
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of Mongersen (GED-0301) for the Treatment of Adult and Adolescent Subjects With Active Crohn's Disease
Brief Title: A Study of Efficacy and Safety of Mongersen (GED-0301) for the Treatment of Adult and Adolescent Subjects With Active Crohn's Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision not to start trial
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GED-0301-CD-003
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; GED-0301; Mongersen; Adolescent; Pediatric; Children
MeSH Terms: conditions — Crohn Disease | interventions — GED0301

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GED-0301 1 x 160 mg once daily (Experimental): GED-0301 1 x 160 mg tablet once daily (QD)
  Interventions: Drug: GED-0301
- GED-0301 - 4 x 40 mg once daily (Experimental): GED-0301 4 x 40 mg tablets once daily (QD)
  Interventions: Drug: GED-0301
- Placebo once daily (Placebo Comparator): Placebo once daily (QD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GED-0301 — GED-0301
  Other Names: Mongersen
  Arms: GED-0301 - 4 x 40 mg once daily; GED-0301 1 x 160 mg once daily
Drug: Placebo — Placebo
  Arms: Placebo once daily

SUMMARY:
The purpose of study is to test the effect of an experimental medication GED-0301(mongersen) and evaluate its safety in patients (≥ 12 years of age) with active Crohn's disease. The study will test GED-0301 compare to placebo for 12 weeks. The study treatment is blinded which means that patients and the study doctor will not know which treatment has been assigned. Patients in this study will be allowed treatment with stable doses of oral aminosalicylates, oral corticosteroids, immunosupressants and antibiotics for the treatment of Crohn's disease. Adolescent patients will also be allowed treatment with stable doses of exclusive enteral nutrition and growth hormone.

All patients who complete the study will have the option to enter a long term active treatment study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

* Male or female ≥ 12 years
* Subject is able to swallow the IP tablets
* Active Crohn's disease (CD) disease as determined by the Crohn's Disease Activity Index (CDAI) score and the Simple Endoscopic Score for Crohn's Disease (SES-CD)
* Must meet a determined average minimum number of daily stools or rating of abdominal pain over a 7day period
* Subject must have failed or experienced intolerance to at least one of the following: budesonide; systemic corticosteroids; immunosuppressants (eg, azathiopurine, 6-mercaptopurine, or methotrexate); or biologics for the treatment of CD (ie, infliximab, adalimumab, certolizumab, or vedolizumab).

Exclusion Criteria:

• The presence of any of the following will exclude a subject from enrollment: Diagnosis of ulcerative colitis (UC), indeterminate colitis, ischemic colitis, microscopic colitis, radiation colitis or diverticular disease-associated colitis, or colitis due to immunodeficiency

* Local manifestations of Crohn's Disease (CD) such as abscesses, short bowel syndrome; or other disease complications for which surgery might be indicated or could confound the evaluation of efficacy
* Subject has strictures with prestenotic dilatation, requiring procedural intervention, or with obstructive symptoms. In addition, subjects with colonic strictures that are not passable with an age-appropriate colonoscope, or strictures in the ileum or ileocecal valve that are fibrotic in nature, will be excluded
* Intestinal resection within 6 months or any intra-abdominal surgery within 3 months prior to the Screening Visit
* Ileostomy or a colostomy
* Subject has a history of any clinically significant medical condition that, in the investigator's opinion, would prevent the subject from participating in the study
* Adolescents with delayed growth or pubertal development who are on corticosteroids at baseline and who should not continue treatment with the same dose of corticosteroids until the Week 12 visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-11-17 (Estimated); Study Completion 2018-12-24 (Estimated)

PRIMARY OUTCOMES:
Clinical remission defined by an average daily liquid or soft stool frequency and abdominal pain score (US) and Crohn's Disease Activity Index (CDAI) (Rest of World) | week 12
  The proportion of subjects achieving clinical remission at Week 12.

SECONDARY OUTCOMES:
Clinical remission defined by an average daily liquid or soft stool frequency and abdominal pain score (US) and CDAI | Week 4, week 12
  The proportion of subjects achieving clinical remission at Week 4, Week 12.
Endoscopic improvement by the Simple Endoscopic Score for Crohn's Disease (SES-CD) | Week 12
  Endoscopic improvement of the mucosa at Week 12.
Clinical response defined by CDAI | Week 4, week 12
  The proportion of subjects achieving clinical response at Week 4, Week 12.
Clinical remission defined by PCDAI | Week 12
  The proportion of subjects achieving clinical remission at Week 12 (adolescent subjects only).
Adverse Events (AEs) | Up to 20 weeks
  Incidence and severity of adverse events
Pharmacokinetics (PK)- plasma concentration of GED-0301 | Week 4, week 8
  The plasma concentration of GED-0301 at Week 4, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Denesh Chitkara, MD, Study Director — Celgene Corporation
Locations (311):
- United States (136):
  - Dcr-Pi Pc, Litchfield Park, Arizona
  - Arizona Digestive Health, Mesa, Arizona
  - Arizona Digestive Health, Phoenix, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Arizona Digestive Health, Sun City, Arizona
  - Gastroenterology Associates PA, Little Rock, Arkansas
  - Valley View Internal Medicine, Garden Grove, California
  - High Desert Gastroenterology, Inc., Lancaster, California
  - University of Southern California Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - Medical Associates Research Group Inc., San Diego, California
  - University of California at San Francisco (PARENT), San Francisco, California
  - HCP Clinical Research LLC, Torrance, California
  - Ventura Clinical Trials, Ventura, California
  - University Of Colorado, Aurora, Colorado
  - Innovative Clinical Research, Lafayette, Colorado
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Medical Research Center of Connecticut LLC, Hamden, Connecticut
  - Connecticut GI PC Research Division, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - University of Miami, Miami, Florida
  - Advance Medical Research Center, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - Sanitas Research, Miami, Florida
  - Galiz Research LLC, Miami Springs, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - GCRM, Orlando, Florida
  - Center For Digestive Health, Orlando, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - East Coast Institute for Research LLC, Saint Augustine, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Cleveland Clinic Florida Weston, Weston, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Georgia Regents University, Augusta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Atlanta Gastroenterology Specialists PC, Suwanee, Georgia
  - Northwestern University-Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University Healthsystem Research Institute, Evanston, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Health Science Research Center, LLC, Pratt, Kansas
  - Heartland Research Associates LLC, Wichita, Kansas
  - Via Christi Research a division of Via Christi Hospitals Wichita Inc, Wichita, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Clinical Trials of SW Louisiana LLC, Lake Charles, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - University of Maryland Medical Group, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Charm City Research Group, Towson, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic Inc. - PARENT ACCOUNT, Burlington, Massachusetts
  - UMass Medical Center, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Medex Research Institute, Caro, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Gastroenterology Associates of Western Michigan PLC, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Mercy Research, Springfield, Missouri
  - Saint Louis University, St Louis, Missouri
  - Mercy Research, Washington, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - AGA Clinical Research Associates LLC, Egg Harbor, New Jersey
  - North Shore-LIJ Health System-Division of Rheumatology, Great Neck, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Montefiore Medical Center PRIME, Lake Success, New York
  - The Feinstein Institute for Medical Research PRIME, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - New York University School of Medicine, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolina Center for Liver Disease, Charlotte, North Carolina
  - Gaffney Health Services, Charlotte, North Carolina
  - PhysiqueMed Clinical Trials, Greensboro, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Clinical Trials of America, LLC, Mount Airy, North Carolina
  - Trial Management Associates LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Ohio Clinical Research Partners LLC, Akron, Ohio
  - Clinical Inquest Center Ltd, Beavercreek, Ohio
  - Dr. Deepak Sarwal, MD, Centerville, Ohio
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Springfield Health Care Center, Springfield, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Main Line Gastroenterology, Havertown, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Penn State University Milton S Hershey Medical Center, State College, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Carolinas Healthcare System, Charleston, South Carolina
  - ClinSearch LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute LLC, Arlington, Texas
  - Gulf Coast Research Group LLC, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Houston Endoscopy and Research Center, Houston, Texas
  - Digestive Health Center, Pasadena, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - University of Utah Division of Gastroenterology, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - University of Virginia, Charlottesville, Virginia
  - Charlottesville Medical Research Center, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Hunter Holmes Mcguire Ctr, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Medical Center Cancer Institute Research, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - The Vancouver Clinic, Vancouver, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Dean Clinic Oregon, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (14):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Centre For Digestive Diseases, Five Dock, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital Institute of Medical and Veterinary Science, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Ballarat Base Hospital, Ballarat
  - Monash Medical Centre Clayton, Bentleigh East
  - St Vincents Hospital Melbourne, Fitzroy
- Austria (3):
  - Klinikum Klagenfurt am Wörtersee, Klagenfurt
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Krankenanstalt Rudolfstiftung Wien, Wein
- Belgium (5):
  - Hopital Universitaire des Enfants, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - CHU Sart Tilman, Liège
- Canada (8):
  - Alberta Childrens Hospital, Calgary, Alberta
  - GI Research Institute, Vancouver, British Columbia
  - Barrie GI Associates, Barrie, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre de sante et de services sociaux Champlain Charles Le Moyne, Greenfield Park, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Clinical Hospital Centre Osijek, Osijek, Croatia
- Czechia (4):
  - Hepato-Gastroenterologie HK, s. r. o., Hradec Králové
  - PreventaMed, Olomouc
  - CCBR Prague CZ, Prague
  - Thomayerova nemocnice, Prague
- Denmark (6):
  - Aarhus Universitetshospital, Aahus C
  - Alborg Universitets Hospital, Aalborg
  - Hvidovre Hospital, Hvidovre
  - Koge Sygehus, Køge
  - Odense Universitetshospital, Odense C
  - Regionshospitalet Silkeborg, Silkeborg
- Finland (2):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Tampereen yliopistollinen sairaala, Tampere
- France (11):
  - CHU Amiens Hopital Sud, Amiens
  - CHU Besancon Hopital Jean Minjoz, Besançon
  - Hopital Claude Huriez CHRU Lille, Lille
  - Hopital Nord CHU Marseille, Marseille
  - CHU Nice Hopital de lArchet 2, Nice
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Reims Hopital Robert Debre, Reims
  - CHU de Rouen Hopital Charles Nicolle, Rouen
  - CHU de Toulouse Hopital Rangueil, Toulouse
  - Hopital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (17):
  - Charite - Campus Virchow-Klinikum, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - St. Josef-Hospital, Bochum
  - Staedisches Klinikum Brandenburg, Brandenburg
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum EssenZentrum fuer Innere Medizin, Essen
  - Kliniken Essen-Mitte, Essen
  - Katholische Kliniken Ruhrhalbinsel GmbH, Essen
  - Crohn Colitis Centrum Rhein Main, Frankfurt
  - Asklepios Klinik Hamburg, Hamburg
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - EUGASTRO GmbH, Leipzig
  - Gastroenterologische Praxis Minden, Minden
  - Universitatsklinikum Regensburg, Regensburg
  - Universitaetsklinikum Ulm, Ulm
  - HELIOS Klinikum Wuppertal, Wuppertal
- Greece (3):
  - General Hospital of Athens Evangelismos, Athens
  - Athens Medical Center, Athens
  - University General Hospital of Patras, Rio Patras
- Hungary (4):
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Szent Margit Korhaz, Budapest
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Szent-Gyorgyi Albert TE AOK Borgyogy, Szeged
- Israel (3):
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (12):
  - Azienda Ospedaliera Universitaria Policlinico Sant Orsola Malpighi, Bologna
  - Fondazione IRCCS CA Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Di Padova, Padua
  - Azienda Ospedaliera Vincenzo Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Universita Campus Bio-Medico di Roma, Roma
  - Complesso Integrato Columbus, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi dAragona, Salerno
  - IRCCS Policlinico San Donato, San Donato Milanese
- Latvia (2):
  - Digestive Diseases Center Gastro, Riga
  - Riga East Clinical University Hospital clinic Gailezers, Riga
- Netherlands (2):
  - Amphia Ziekenhuis, Breda
  - Erasmus Medisch Centrum, Rotterdam
- Poland (6):
  - SP ZOZ Wojewodzki Szpital Zespolony im. J. Sniadeckiego, Bialystok
  - Clinsante S.C. Osrodek Badan Klinicznych, Bydgoszcz
  - Centrum Medyczne A-Z Clinic, Krakow
  - Centrum Medyczne AMED, Lodz
  - Nzoz Vivamed, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
- Portugal (5):
  - Hospital de Braga, Braga
  - Hospital da Senhora da Oliveira Guimaraes, Guimarães
  - Hospital Da Luz, Lisbon
  - Centro Hospitalar de Sao Joao, EPE, Porto
  - Centro Hospitalar do Alto Minho - Unidade Local de Saúde do Alto Minho, EPE, Viana do Castelo
- Romania (2):
  - CMI Dr. Tirnaveanu Amelita, Oradea
  - Centrul de Gastroenterologie Dr. Goldis, Timișoara
- Russia (5):
  - Medical Center Stolitsa-Medikl, Moscow
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - FSBI Scientific Research Institute of Physyology and Basic Medicine under the SB of RAMS, Novosibirsk
  - SPb SBIH City Hospital # 26, Saint Petersburg
  - NonState Healthcare Institution Central Clinical Hospital, Samara station JSC Russian Railways, Samara
- Clinical Center Bezanijska Kosa, Belgrade, Serbia
- GASTRO I., s.r.o., Prešov, Slovakia
- South Korea (11):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Hanyang Univerisy Guri Hospital, Guri-si
  - CHA Bundang Medical Center CHA University, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (9):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de la Princessa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario Miguel Servet, Zaragoza
- Danderyds Sjukhus AB, Stockholm, Sweden
- Switzerland (4):
  - Inselspital - Universitaetsspital Bern, Bern
  - Crohn-Colitis Zentrum Bern Gemeinschaftspraxis Balsiger Seibold und Partner, Bern
  - Hopitaux Universitaires de Geneve-HUG, Geneva
  - UniversitatSspital Zurich, Zurich
- Turkey (Türkiye) (15):
  - Ankara University Medical Faculty, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Turkiye Yuksek Ihtisas Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Firat University Medical Faculty, Elâzığ
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Acibadem Fulya Hospital, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Istanbul Medeniyet Uni Goztepe Training&Res Hosp, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Izmir, Izmir
  - Kocaeli Derince Training and Research Hospital, Kocaeli
  - Inonu Uni. Med. Fac., Malatya
  - Mersin University Medical Faculty, Mersin
- Ukraine (9):
  - CI of PH Kharkiv CCH #2, Kharkiv
  - Treatment-Diagnostic Center of Private Enterprise of PMF Atsynus, Kirovohrad
  - Kyiv City Clinical Hospital #1, Kyiv
  - CI Odesa Regional Clinical Hospital, Odesa
  - CI of SRC Sumy RCH Dept of Rheumatology Sumy SU MI, Sumy
  - Ternopil City Communal Emergency Medical Care Hospital, Ternopil
  - SRI of Invalid Rehabilitation EST Complex of Vinnytsia M.I.Pyrogov NMU MOHU, Vinnytsia
  - SI Branch CH of Zaporizhzhia Station-2 of SE Prydniprovska Railway Dept of Surgery Zaporizhzhia SMU, Zaporizhia
  - CI Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhya
- United Kingdom (9):
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - University Hospital Coventry, Coventry
  - Queen Elizabeth University Hospital, Glasgow
  - Hull Royal Infirmary, Hull
  - Royal London Hospital, London
  - University College London Hospitals, London
  - Manchester Royal Infirmary, Manchester
  - Nottingham University Hospitals Queens Medical Centre, Nottingham
  - Borders General Hospital, Roxburghshire